CLINICAL TRIAL: NCT02458937
Title: Functional Outcomes for Children, Adolescents, and Young Adults With Osteonecrosis Following Hip Core Decompression
Brief Title: Functional Outcomes Following Hip Core Decompression in Younger Participants With Osteonecrosis
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Tennessee Physical Therapy Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: ONFUNC
Record Dates: First submitted 2015-05-13; First posted 2015-06-01 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Osteonecrosis
Keywords: Leukemia; Hodgkin Disease; Non-Hodgkin's Lymphoma; Sickle Cell Disease; Hip Core Decompression; Function Outcomes
MeSH Terms: conditions — Osteonecrosis; Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Anemia, Sickle Cell | interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteonecrosis: Observational measures of functional outcomes will be obtained from all participants who consent to and complete the study.
  Interventions: Functional Mobility Assessment (FMA), GAITRite® System, and Range of Motion.
  Interventions: Other: Functional Mobility Assessment; Other: GAITRite® System; Other: Range of Motion

INTERVENTIONS:
Other: Functional Mobility Assessment — Functional Mobility Assessment (FMA) is a tool that was developed to measure functional mobility in children and adolescents with lower-extremity sarcoma. It is comprised of well-established outcome measures that examine various domains of function. The six categories tested by the FMA include pain, functional mobility, use of assistive devices, satisfaction with quality of gait, participation in the community, and endurance.
  Other Names: FMA
Other: GAITRite® System — Subjects will be required to walk at a self-selected comfortable pace and again at fast speed. Software will then calculate and report the temporo-spatial gait parameters for collection and evaluation by the primary investigator.
  Other Names: Portable Walkway
Other: Range of Motion — Measurements will include hip flexion, hip abduction and adduction, and hip internal and external rotation. Range of motion (ROM) will be attempted on bilateral lower extremities, however if post-operative ROM precautions are implemented, the involved extremity will not be measured. Goniometry is a reliable and valid measure for active and passive ROM when following standardized procedures.
  Other Names: Goniometer; ROM

SUMMARY:
Although uncommon in the general pediatric population, osteonecrosis (ON) is prevalent in children and adolescents with cancer, particularly among those that have had chronic exposure to glucocorticoids and among those having undergone allogeneic hematopoietic stem cell transplantation. Patients with hematologic disease are also at risk for developing ON.

Hip Core Decompression (HCD) is a widely used surgical procedure with several studies reporting positive results; however, most are subject to criticism because of the limited sample size or the absence of appropriate functional outcome measures.

The objective of this pilot study is to observe and collect information on several functional outcome measures and assess if Hip Core Decompression (HCD) potentially improves functional outcomes in children, adolescents and young adults with osteonecrosis.

PRIMARY OBJECTIVE:

* To describe functional outcomes of children, adolescents, and young adults with osteonecrosis of the femoral head following hip core decompression surgery. Parameters assessed will include pain, functional mobility, endurance, quality of life, and gait patterns pre-operatively and post-operatively over time.

DETAILED DESCRIPTION:
Hip core decompression (HCD) is not being done as part of this study. Rather, patients who are undergoing HCD at St. Jude Children's Research Hospital (SJCRH) will be observed for functional outcomes following the procedure.

HCD is considered an excellent surgical option when considering the multiple issues among this population, which include young age, the natural progression of osteonecrosis to femoral head collapse, the limited life expectancy of the prosthetic technology currently available for total hip arthroplasty (THA), and patient quality of life. This study will seek to describe functional outcomes and quality of gait following HCD in a pediatric population with osteonecrosis. The results of this study will provide valuable information as to the functional limitations within this population pre- and post-operatively.

For each research participant the observations on all outcome measures of interest will be collected at 5 time points: pre-operatively (baseline measure), and post-operatively at 6 weeks, 12 weeks, 6 months and 1 year. These time points will allow for comparison between pre- and post-operative outcomes to determine if outcomes are improved following surgery, and if these outcomes continue to improve over time. This study will also provide a foundation for the future development of treatment programs designed to target identified limitations specific to this population.

ELIGIBILITY:
Inclusion Criteria:

* Patient being treated at St. Jude Children's Research Hospital
* Diagnosis of osteonecrosis of the hip
* Diagnosis of hematologic malignancy or sickle cell disease
* Age between 8 and 29 years of age
* Patient and/or parent or legal guardian must sign a written informed consent
* Patient is considered an acceptable candidate for hip core decompression surgery by his/her primary physician and orthopedic surgeon

Exclusion Criteria:

* Patient with a diagnosis that is not a hematologic malignancy or sickle cell disease
* Patient that has had amputation or reconstructive surgery of the lower extremities
* Premorbid condition that prevents patient from ambulating
* Patient that has a serious, non-healing wound, ulcer, or bone fracture

Ages: 8 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be patients with osteonecrosis at St. Jude Children's Research Hospital who receive hip core decompression surgery as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Degree of Pain | At 1 year after surgery
  Pain is measured by using a numeric scale requiring patients to rate any pain experienced in the prior week on a 0 (no pain) to 10 (worst pain imaginable) scale
Functional Mobility | At 1 year after surgery
  Functional mobility will be measured by using the Timed Up and Down Stairs (TUDS) and Timed Up and Go (TUG). TUDS assesses the time required for a patient to walk up and down 12 stairs to measure functional mobility, balance, and motor skills. TUG measures the time needed to stand from a seated position, ambulate 3 meters, turn around, return to chair and resume sitting. This will provide a measure of dynamic balance and mobility.
Physiological Cost Index (PCI) | At 1 year after surgery
  Endurance will be assessed following completion of the 9-Minute Run-Walk Test. The patient will be instructed to walk or run for 9 minutes while trying to cover as much distance as possible. Heart rate (HR) and rate of perceived exertion (RPE) data will be collected during the walk/run. RPE measures the level of the patient's exertion using a likert scale of numbers (6-20) and adjectives describing effort. A wheeled feet counter will measure distance and a stopwatch will track time. Upon completion of the 9-minute run-walk, the physiological cost index (PCI) will be calculated by dividing the difference in the patient's heart rate (HR while walking- HR at rest) by walking speed in meters per minute.
Quality of Life | At 1 year after surgery
  The use of supports, patient satisfaction, and participation in the community will be measured by patient provided responses to questions pertaining to the use of supports (brace, cane, crutches), satisfaction with walking quality, and participation in school, work, and/or sports. The responses will be scored on a 0-5 scale, with 0 demonstrating the least preferred outcome.
Temporo-Spatial Gait Parameters | At 1 year after surgery
  Subjects will be required to walk at a self-selected comfortable pace and again at fast speed. Software will then calculate and report the temporo-spatial gait parameters for collection and evaluation by the primary investigator.
Range of Motion | At 1 year after surgery
  Active and passive ROM will be measured using a goniometer. Measurements will include hip flexion, hip abduction and adduction, and hip internal and external rotation. ROM will be attempted on bilateral lower extremities, however if post-operative ROM precautions are implemented, the involved extremity will not be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M. DeFeo, PT, DPT, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols